CLINICAL TRIAL: NCT02959203
Title: Comparison of Bedside Ultrasound With Chest X-ray to Detect CVC Related Mechanical Complications; a Prospective Observational Study (COMBUX-study)
Brief Title: Comparison of Bedside Ultrasound With Chest X-ray for Confirmation of Central Venous Catheter Position
Acronym: COMBUX
Status: Completed | Type: Observational
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Groene Hart Ziekenhuis (Other)
Responsible Party: Principal Investigator, Jasper Smit, BSc, Amsterdam UMC, location VUmc
Other Study IDs: 2016.053
Record Dates: First submitted 2016-11-04; First posted 2016-11-09 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Pneumothorax Iatrogenic Postprocedural; Malposition, Central Venous Catheter
Keywords: Central Venous Catheter; Ultrasound; Chest X-ray; Pneumothorax
MeSH Terms: conditions — Pneumothorax

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Background:

Insertion of a central venous catheter (CVC) could lead to a variety of complications.

To detect those complications, Chest X-ray (CXR) is still the reference standard. However, there are major limitations in performing CXR's in the critical care setting.

Aim/objectives:

The objective of this study is to compare the use of bedside ultrasound (US) to conventional CXR in visualization of accuracy and safety of the CVC placement. The aim is to eventually replace X-ray with bedside ultrasound as gold standard for the confirmation of CVC-placement in critically ill patients, thereby reducing radiation exposure and unnecessary delay before CVC use.

Methods:

The bedside US will be performed by the student or attending physician, who is blinded for CXR findings. After US examination, the attending physician (or student) will fill in a structured form, based on an established protocol. CXR will be performed before or after US examination and assessed by a radiologist. The radiologist will be blinded for the findings of the bedside ultrasound to prevent any biases. Final diagnosis will be determined after examination of the complete medical chart.

DETAILED DESCRIPTION:
Most patients admitted to an intensive care unit undergo central venous catheterization (CVC) or already have received a CVC. Over 5 million CVC placements are performed each year in the United States. An indication of central venous access is for example when peripheral veins are inaccessible or for the administration of potent vasoactive drugs such as norepinephrine or dopamine. Three anatomical sites are frequently used to insert a CVC: the subclavian, jugular and femoral site. Although central venous catheterization offers multiple advantages, it is associated with adverse events that could be hazardous for patients. Mechanical, infectious or thrombotic complications could occur. Most common mechanical complications include arterial puncture, hematoma and pneumothorax. Besides mechanical complications, malposition of a CVC could also lead to complications, including phlebitis, perforation, and venous thrombosis or occlusion. Malposition of the CVC tip into the right atrium could also lead to arrhythmias. The frequency of primary mal-positioning has been shown to be up to 3.7%. A recent multicenter trial, which included 3471 catheters in 3027 patients, showed that subclavian-vein catheterization was associated with a lower risk of bloodstream infection and symptomatic thrombosis but involved a higher risk of pneumothorax as compared to jugular-vein or femoral-vein catheterization. The risk of mechanical complications in subclavian, jugular or femoral catheterization was 2.1%, 1.4% and 6% respectively.

To date, the post-procedural chest X-ray (CXR) has been the reference standard to detect these mechanical complications. Some studies suggest that it should not be considered a reliable procedure for detecting complications in the absence of clinical symptoms. In addition, reading of a bedside CXR alone is not very accurate to identify intra-atrial tip position. The exceedingly low complication rate after right internal jugular vein catheterization suggests that, to detect pneumothorax and intra-atrial malposition, routine post-procedure CXR is neither necessary nor accurate and causes delay until catheter use. Omitting the need for CXR could reduce healthcare costs as well.

Due to some clear advantages, there has already been an increasing role for ultrasonography in the critical care setting. In comparison to radiography, an advantage of ultrasound is that the patient is not exposed to radiation, and is often faster performed. Compared to the traditional 'blind' landmark method, ultrasound-guided subclavian cannulation reduces failed catheterizations and complications associated with subclavian catheterization. Advantages of ultrasound-guided cannulation include correct identification of the vein, detecting variable anatomy and reducing events of arterial puncture. Due to the developing knowledge and techniques in ultrasound, is has been suggested that it would be a suitable method to replace CXR in the role of detecting pneumothorax and identifying CVC tip position. A small number of studies already demonstrated this effect.

In this study we evaluate the use of ultrasound as diagnostic modality in patients after CVC placement in the subclavian or jugular vein. This research proposal aims to evaluate US examination as diagnostic tool for misplacement, bleeding and pneumothorax after CVC-placement. Combining the different strategies from previous studies. we developed "tHe UltraSound evaluation of Cvc Insertion" i.e. HUSCI-protocol. Hereby, we aim to improve accuracy The outcome measure will be the sensitivity and specificity of US. In addition, diagnostic concordance between US and CXR in patients after CVC placement will be studied. If US catches clinical relevant findings accurately we can replace standard expensive and harmful CXR as standard diagnostic tool in patients after CVC-placement in the future. We hypothesize that US can confirm correct CVC placement and detect potential associated complications accurately.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18
* Central venous cannulation performed
* CVC in internal jugular vein or subclavian vein

Exclusion Criteria:

* Refusal to undergo ultrasound examination
* Refusal to undergo chest X-ray
* CVC in femoral vein
* PICC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who undergo central venous cannulation
Sampling Method: Non-Probability Sample
Enrollment: 750 (Actual)
Dates: Start 2016-06; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of ultrasound to detect CVC malposition | Accuracy will be measured after ultrasound and Chest X-ray evaluation (expected time frame: 3 hours)
  Sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV) are used as accuracy outcome parameters. A 'true positive' result is defined as an US-suggested aberrant position of the CVC (catheter tip in any other vein than the superior vena cava (SVC), outside the venous system, or positioned deep in the right atrium or ventricle) confirmed by CXR. If bedside US rules out an aberrant position of the catheter tip correctly it is considered to be a 'true negative' result

SECONDARY OUTCOMES:
Feasibility of ultrasound | Feasiblity will be measured after ultrasound and Chest X-ray evaluation (expected time frame: 3 hours)
  Ultrasound is considered to be feasible if all US-views in the protocol can be obtained
Diagnostic accuracy of ultrasound to detect pneumothorax | Accuracy will be measured after ultrasound and Chest X-ray evaluation (expected time frame: 3 hours)
  Interobserver and overall percent agreement between US and CXR is calculated

CONTACTS AND LOCATIONS:
Locations (1):
- VU University Medical Center, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hourmozdi JJ, Markin A, Johnson B, Fleming PR, Miller JB. Routine Chest Radiography Is Not Necessary After Ultrasound-Guided Right Internal Jugular Vein Catheterization. Crit Care Med. 2016 Sep;44(9):e804-8. doi: 10.1097/CCM.0000000000001737. PMID 27035241
- [Background] Lalu MM, Fayad A, Ahmed O, Bryson GL, Fergusson DA, Barron CC, Sullivan P, Thompson C; Canadian Perioperative Anesthesia Clinical Trials Group. Ultrasound-Guided Subclavian Vein Catheterization: A Systematic Review and Meta-Analysis. Crit Care Med. 2015 Jul;43(7):1498-507. doi: 10.1097/CCM.0000000000000973. PMID 25803646
- [Background] Lichtenstein D, van Hooland S, Elbers P, Malbrain ML. Ten good reasons to practice ultrasound in critical care. Anaesthesiol Intensive Ther. 2014 Nov-Dec;46(5):323-35. doi: 10.5603/AIT.2014.0056. PMID 25432552
- [Background] Parienti JJ, Mongardon N, Megarbane B, Mira JP, Kalfon P, Gros A, Marque S, Thuong M, Pottier V, Ramakers M, Savary B, Seguin A, Valette X, Terzi N, Sauneuf B, Cattoir V, Mermel LA, du Cheyron D; 3SITES Study Group. Intravascular Complications of Central Venous Catheterization by Insertion Site. N Engl J Med. 2015 Sep 24;373(13):1220-9. doi: 10.1056/NEJMoa1500964. PMID 26398070
- [Background] Zadeh MK, Shirvani A. The role of routine chest radiography for detecting complications after central venous catheter insertion. Saudi J Kidney Dis Transpl. 2014 Sep;25(5):1011-6. doi: 10.4103/1319-2442.139895. PMID 25193899
- [Background] Vezzani A, Manca T, Vercelli A, Braghieri A, Magnacavallo A. Ultrasonography as a guide during vascular access procedures and in the diagnosis of complications. J Ultrasound. 2013 Oct 29;16(4):161-70. doi: 10.1007/s40477-013-0046-5. eCollection 2013 Oct 29. PMID 24432170
- [Background] Nayeemuddin M, Pherwani AD, Asquith JR. Imaging and management of complications of central venous catheters. Clin Radiol. 2013 May;68(5):529-44. doi: 10.1016/j.crad.2012.10.013. Epub 2013 Feb 13. PMID 23415017
- [Background] Wirsing M, Schummer C, Neumann R, Steenbeck J, Schmidt P, Schummer W. Is traditional reading of the bedside chest radiograph appropriate to detect intraatrial central venous catheter position? Chest. 2008 Sep;134(3):527-533. doi: 10.1378/chest.07-2687. Epub 2008 Jul 18. PMID 18641117
- [Background] Taylor RW, Palagiri AV. Central venous catheterization. Crit Care Med. 2007 May;35(5):1390-6. doi: 10.1097/01.CCM.0000260241.80346.1B. PMID 17414086
- [Background] McGee DC, Gould MK. Preventing complications of central venous catheterization. N Engl J Med. 2003 Mar 20;348(12):1123-33. doi: 10.1056/NEJMra011883. No abstract available. PMID 12646670
- [Background] Bedel J, Vallee F, Mari A, Riu B, Planquette B, Geeraerts T, Genestal M, Minville V, Fourcade O. Guidewire localization by transthoracic echocardiography during central venous catheter insertion: a periprocedural method to evaluate catheter placement. Intensive Care Med. 2013 Nov;39(11):1932-7. doi: 10.1007/s00134-013-3097-3. Epub 2013 Sep 20. PMID 24052186
- [Background] Cortellaro F, Mellace L, Paglia S, Costantino G, Sher S, Coen D. Contrast enhanced ultrasound vs chest x-ray to determine correct central venous catheter position. Am J Emerg Med. 2014 Jan;32(1):78-81. doi: 10.1016/j.ajem.2013.10.001. Epub 2013 Oct 9. PMID 24184012
- [Background] Vezzani A, Brusasco C, Palermo S, Launo C, Mergoni M, Corradi F. Ultrasound localization of central vein catheter and detection of postprocedural pneumothorax: an alternative to chest radiography. Crit Care Med. 2010 Feb;38(2):533-8. doi: 10.1097/CCM.0b013e3181c0328f. PMID 19829102
- [Background] Gekle R, Dubensky L, Haddad S, Bramante R, Cirilli A, Catlin T, Patel G, D'Amore J, Slesinger TL, Raio C, Modayil V, Nelson M. Saline Flush Test: Can Bedside Sonography Replace Conventional Radiography for Confirmation of Above-the-Diaphragm Central Venous Catheter Placement? J Ultrasound Med. 2015 Jul;34(7):1295-9. doi: 10.7863/ultra.34.7.1295. PMID 26112633
- [Background] Kim SC, Graff I, Sommer A, Hoeft A, Weber S. Ultrasound-guided supraclavicular central venous catheter tip positioning via the right subclavian vein using a microconvex probe. J Vasc Access. 2016 Sep 21;17(5):435-9. doi: 10.5301/jva.5000518. Epub 2016 Mar 22. PMID 27012271
- [Background] Maury E, Guglielminotti J, Alzieu M, Guidet B, Offenstadt G. Ultrasonic examination: an alternative to chest radiography after central venous catheter insertion? Am J Respir Crit Care Med. 2001 Aug 1;164(3):403-5. doi: 10.1164/ajrccm.164.3.2009042. PMID 11500340